CLINICAL TRIAL: NCT03777332
Title: A 24-Month Phase Ib Multi-Center, Open Label, Single Arm Study to Evaluate the Safety of Intravitreal APL-2 Therapy in Patients Diagnosed With Geographic Atrophy (GA) Secondary to Age-Related Macular Degeneration (AMD)
Brief Title: Study to Evaluate the Safety of Intravitreal APL-2 in Patients Diagnosed With Geographic Atrophy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL2-103
Record Dates: First submitted 2018-12-14; First posted 2018-12-17 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Geographic Atrophy
MeSH Terms: conditions — Geographic Atrophy | interventions — pegcetacoplan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- (Cohort 1) Pegcetacoplan, 15 mg/100 μL, monthly for up to 60 months (Experimental)
  Interventions: Drug: PEGCETACOPLAN (APL-2)
- (Cohort 2) Pegcetacoplan, 15 mg/100 μL, monthly for up to 36 months (Experimental)
  Interventions: Drug: PEGCETACOPLAN (APL-2)
- (Cohort 2) Pegcetacoplan, 15 mg/100 μL, every other month for up to 36 months (Experimental)
  Interventions: Drug: PEGCETACOPLAN (APL-2)

INTERVENTIONS:
Drug: PEGCETACOPLAN (APL-2) — Complement (C3) Inhibitor

SUMMARY:
Safety Assessment of APL-2 in Patients with Geographic Atrophy

ELIGIBILITY:
Inclusion Criteria: Cohort 1

The study eye must meet all inclusion criteria. If both eyes meet the inclusion criteria, the eye with the worst normal luminance best-corrected visual acuity (NL-BCVA) at the screening visit will be designated as the study eye. If both eyes have the same visual acuity, the eye with the larger GA lesion will be selected as the study eye. If both eyes have the same GA lesion size, the right eye will be selected as the study eye.

Ocular- specific inclusion criteria apply to the study eye only, unless otherwise specified.

1. Age ≥ 60 years.
2. Normal Luminance best corrected visual acuity of between 35 and 5 letters using Early Treatment Diabetic Retinopathy Study (ETDRS) charts (approximately between 20/200 and 20/800 Snellen equivalent).
3. Clinical diagnosis of GA of the macula secondary to AMD as determined by the Investigator and confirmed by the Reading Center.
4. The GA lesion must meet the following criteria as determined by the central reading center's assessment of Fundus Autofluorescence (FAF) imaging at screening:

   1. Total GA area must be ≥ 2.5 (1 disk areas [DA]).
   2. If GA is multifocal, at least one focal lesion must be ≥ 1.25 mm2 (0.5 DA), with the overall aggregate area of GA as specified above in 4a.
5. Adequate clarity of ocular media, adequate pupillary dilation, and fixation to permit the collection of good quality images as determined by the Investigator.
6. Female subjects must be:

   1. Women of non-child-bearing potential (WONCBP), or
   2. Women of child-bearing potential (WOCBP) with a negative serum pregnancy test at screening and must agree to use protocol defined methods of contraception for the duration of the study and refrain from breastfeeding for the duration of the study.
7. Males with female partners of child-bearing potential must agree to use protocol defined methods of contraception and agree to refrain from donating sperm for the duration of the study.
8. Willing and able to give informed consent and to comply with the study procedures and assessments.

Exclusion Criteria: Cohort 1

Ocular specific exclusion criteria apply to the study eye only, unless otherwise specified.

1. GA secondary to a condition other than AMD such as Stargardt disease, cone rod dystrophy or toxic maculopathies like plaquenil maculopathy in either eye.
2. Spherical equivalent of the refractive error demonstrating > 6 diopters of myopia or an axial length >26 mm.
3. Any history or active choroidal neovascularization (CNV), associated with AMD or any other cause, including any evidence of retinal pigment epithelium rips or evidence of neovascularization anywhere based on SD-OCT imaging and/or fluorescein angiography as assessed by the Reading Center.
4. Presence of an active ocular disease that in the opinion of the Investigator compromises or confounds visual function, including but not limited to, uveitis, other macular diseases (e.g. clinically significant epiretinal membrane [ERM], full thickness macular hole) or uncontrolled glaucoma/ocular hypertension). Benign conditions in the opinion of the Investigator such as peripheral retina dystrophy are not exclusionary.
5. Intraocular surgery (including lens replacement surgery) within 3 months prior to enrollment.
6. History of laser therapy in the macular region.
7. History of intraocular injection within 3 months prior to the screening visit.
8. Aphakia or absence of the posterior capsule. Note: Yttrium-Aluminum Garnet YAG laser posterior capsulotomy for posterior capsule opacification done at least 60 days prior to screening is not exclusionary.
9. Any ocular condition other than GA secondary to AMD that may require surgery or medical intervention during the study period or, in the opinion of the Investigator, could compromise visual function during the study period.
10. Any contraindication to IVT injection including current ocular or periocular infection.
11. Participation in any systemic experimental treatment or any other systemic investigational new drug including within 6 weeks or 5 half-lives of the active ingredient (whichever is longer) prior to the start of study treatment. Note: clinical trials solely involving observation, over-the-counter vitamins, supplements, or diets are not exclusionary.
12. Medical or psychiatric conditions that, in the opinion of the Investigator, make consistent follow-up over the 60-month treatment period unlikely, or would make the subject an unsafe study candidate.
13. Any screening laboratory value (hematology, serum chemistry or urinalysis) that in the opinion of the Investigator is clinically significant and not suitable for study participation.
14. Known hypersensitivity to fluorescein sodium for injection or hypersensitivity to pegcetacoplan or any of the excipients in pegcetacoplan solution.

Inclusion Criteria: Cohort 2

Ocular-specific inclusion criteria apply to the study eye only.

1. Participated in the APL2-303 (Derby, NCT03525613) or APL2-304 (Oaks, NCT03525600) study with completion of the Month 24 visit and have been invited to participate in this study.

   a. Subjects who did not discontinue treatment but missed the Month 24 visit are also eligible to participate in this study.
2. Clarity of ocular media, adequate pupillary dilation, and fixation to permit the collection of good quality images as determined by the investigator.
3. Female subjects must be:

   1. Women of non-child-bearing potential (WONCBP), or
   2. Women of child-bearing potential (WOCBP) with a negative serum pregnancy test at screening and must agree to use protocol defined methods of contraception for the duration of the study and 90 days after their last dose of pegcetacoplan, and refrain from breastfeeding for the duration of the study.
4. Males with female partners of child-bearing potential must agree to use protocol defined methods of contraception and agree to refrain from donating sperm for the duration of the study and for 90 days after their last dose of pegcetacoplan.
5. Willing and able to give informed consent to comply with the study procedures and assessments

Exclusion Criteria: Cohort 2

Ocular-specific exclusion criteria apply to the study eye only, unless otherwise specified.

1. Subjects who discontinued the study drug prior to Month 24 and remained in the APL2- 303 (Derby, NCT 03525613) or APL2-304 (Oaks, NCT03525600 study for safety assessments. Temporary pause of the study drug is not exclusionary.
2. Presence of an active ocular disease that, in the opinion of the investigator, compromises or confounds visual function, including, but not limited to, macular hole or other macular diseases (eg, clinically significant epiretinal membrane). Benign conditions in the opinion of the investigator such as peripheral retinal dystrophy are not exclusionary.
3. Any contraindication to IVT injection including current ocular or periocular infection.
4. Medical or psychiatric conditions that, in the opinion of the investigator, is clinically significant and not suitable for study participation or consistent follow-up.
5. Known hypersensitivity to fluorescein sodium for injection or hypersensitivity to pegcetacoplan or any of the excipients in pegcetacoplan solution.
6. Pregnancy, breastfeeding, or positive pregnancy test.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Ocular and Systemic Treatment-Emergent Adverse Events (TEAEs) | 25 Months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - California Retina Consultants, Bakersfield, California
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - The Retina Partners, Encino, California
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Retina Consultants of Houston, The Woodlands, Texas

REFERENCES:
- [Derived] Wykoff CC, Holz FG, Chiang A, Boyer D, Dhoot DS, Loewenstein A, Mones J, Heier J, Abbey AM, Singerman LJ, Vajzovic L, Lin J, Li C, Vilupuru A, Baumal CR; OAKS, DERBY, and GALE Investigators. Pegcetacoplan Treatment for Geographic Atrophy in Age-Related Macular Degeneration Over 36 Months: Data From OAKS, DERBY, and GALE. Am J Ophthalmol. 2025 Aug;276:350-364. doi: 10.1016/j.ajo.2025.04.016. Epub 2025 Apr 23. PMID 40280279